CLINICAL TRIAL: NCT00675558
Title: Bariatric Surgery for Morbid Obesity: Clinical and Pathophysiologic Consequences
Brief Title: Bariatric Surgery for Morbid Obesity
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Paul D. Berk, Professor, Department of Medicine, Digestive & Liver Diseases, Columbia University
Other Study IDs: AAAC0355; R01DK072526 (NIH)
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Obesity; Morbid Obesity
Keywords: Obesity; morbid obesity; bariatric surgery
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and biopsies of omental and subcutaneous fat.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-Obese (NO): Patients with a BMI < 29.9 scheduled for clinically indicated laparoscopic abdominal surgery.
  Interventions: Procedure: Initial Surgery
- Morbidly Obese (MO): Patients with a BMI > 40.0 scheduled for clinically indicated laparoscopic abdominal surgery.
  Interventions: Procedure: Initial Surgery
- Super-morbidly Obese (SMO): Patients with a BMI > 50.0 scheduled for clinically indicated laparoscopic abdominal surgery.
  10 subjects of the original 30 subjects enrolled into this group received a second bariatric procedure. The remaining 20 subjects of the original 30 subjects did not continue on to the second phase (second bariatric surgery) of the study.
  Interventions: Procedure: Initial Surgery; Procedure: Second Bariatric Surgery

INTERVENTIONS:
Procedure: Initial Surgery — NO patients had initial abdominal laparoscopic surgery at study entry, during which research fat biopsies were obtained, completing their participation.
  MO patients had initial laparoscopic bariatric surgery (gastric bypass, adjustable gastric band, or sleeve gastrectomy) and fat biopsies at entry, completing their participation.
  All 30 SMO patients had initial laparoscopic bariatric surgery (sleeve gastrectomy) & fat biopsies. The first 10 to lose 100 lbs but who needed further surgery to reach optimal weight and who consented to further surgery underwent a 2nd laparoscopic bariatric surgery (either a biliopancreatic diversion with duodenal switch or a Roux-en-Y gastric bypass) and biopsies. The interval between surgeries averaged 15 mos. and the weight loss 55 kg. 30 SMO patients were initially enrolled to insure that 10 would complete 2 surgeries. When 10 had had their 2nd operation, the study was considered complete, and the remaining 20 SMO participants were so notified.
  Other Names: Intervention names:; NO patients all had one surgery: Abdominal Laparoscopic Surgery. Specific procedure determined by underlying medical condition.; MO patients all had one surgery: Abdominal Laparoscopic Bariatric Surgery.; All 30 SO patients had an initial Abdominal Laparoscopic Bariatric Surgery.; The first 10 SMO patients to meet defined requirements had a second Abdominal Laparoscopic Bariatric Surgery. Details below.
Procedure: Second Bariatric Surgery — A second bariatric procedure was performed on only 10 of the original 30 Super-morbidly Obese (SMO) subjects.
  Groups: Super-morbidly Obese (SMO)

SUMMARY:
Despite progress in understanding the pathophysiology of obesity, current strategies for its medical management remain largely ineffective. Most efforts have focused on reducing caloric intake or increasing energy expenditure, either through behavior modification (e.g. dieting, regular exercise) alone, or augmented by pharmacologic efforts to decrease appetite, inhibit fat absorption, or alter metabolism. Bariatric surgery remains the only proven long term treatment of morbid obesity.

Super morbidly obese (SMO: Body Mass Index (BMI) > 50) and super super morbidly obese (SSMO: BMI > 60) patients lose considerable weight, but stabilize at Body Mass Indexes (BMIs) that are still obese or even morbidly obese after risking considerable morbidity and/or mortality. Among commonly performed bariatric surgeries, a laparoscopic two-stage procedure, in which an initial restrictive procedure is followed after a weight loss of ~100 lbs by a more complex procedure that creates malabsorption, is gaining interest. Initial studies have demonstrated very good long-term weight loss with minimal morbidity, and no operative mortality in these high risk patients.

Availability of biospecimens obtained at each stage of this protocol will allow participating scientists a unique opportunity to test in human tissues hypotheses developed in animals. Studies proposed under this application focus on fatty acids and overall fat disposition in fat depots (adipose tissue) of your body, and the role of adipose tissue hormones and inflammatory processes in obesity and its associated health related issues.

DETAILED DESCRIPTION:
Despite rapidly growing interest in the pathogenesis of the obesity epidemic, the pathophysiology of obesity remain poorly understood. While studies in animals have yielded many insights, it has become clear that human obesity differs in important ways from that in rodents. Bariatric surgery offers better outcomes, but in the highest grades of obesity (BMI>50) remains a high risk undertaking with >5% operative mortality being reported when commonly performed bariatric surgical approaches are employed. By contrast, laparoscopic two-stage approach has resulted in excellent weight loss, minimal morbidity, and <1% mortality.

Availability of blood samples and biopsies of omental and subcutaneous fat from each of the paired bariatric procedures in this protocol will provide a unique opportunity to study key issues in human obesity. This study tests the broad hypothesis that there are significant and as yet unrecognized differences between the pathobiology of obesity in man and rodents, the identification of which may lead to new therapeutic targets. Accordingly, to facilitate comparisons with aspects of obesity we have already investigated in animal models, we will 1. seek fat depot specific differences in Long Chain Fatty Acid (LCFA) disposition, macrophage infiltration and adipokine production in obesity and after surgery-induced weight loss in man, and correlate them with the presence/severity of the metabolic syndrome (MetSyn); and 2., quantify the relative significance and response to weight loss of different mechanisms contributing to hepatic steatosis and the elevated triglycerides (TG) and reduced High-Density Lipoprotein (HDL) typical of obesity and MetSyn.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 - 75 years of age
* Scheduled to have two stage bariatric surgery
* BMI > 50

Exclusion Criteria:

* Younger than 18 or older than 75 years of age
* Underlying cardiac disease or other medical condition that increases the risk of their surgical procedure
* Pregnancy
* Sufficiently diminished mental capacity so as to be unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will be drawn from adults referred for bariatric surgery at New York Presbyterian Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2011-04 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Berk, M.D, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients referred to several Divisions of the Department of Surgery at New York Presbyterian Hospital.
Groups:
- Super-morbidly Obese (SMO): Patients with a BMI > 50.0 scheduled for clinically indicated laparoscopic abdominal surgery.
  10 subjects of the original 30 subjects enrolled into this group received a second bariatric procedure. The remaining 20 subjects of the original 30 subjects did not continue on to the second phase (initial bariatric surgery) of the study.
Period: Surgery
Arm/Group | Non-Obese (NO) | Morbidly Obese (MO) | Super-morbidly Obese (SMO)
Started | 10 | 10 | 30
Completed | 10 | 10 | 30
Not Completed | 0 | 0 | 0
Period: Second Operation
Arm/Group | Non-Obese (NO) | Morbidly Obese (MO) | Super-morbidly Obese (SMO)
Started | 0 (No medical reason, and no study-related reason for non-obese pts to have a second procedure.) | 0 (No medical reason, and none for the goals of the study, for MO pts to have a second procedure .) | 10 (As predicted, only 10 SMO patients medically required a second operation, and thus met study goals.)
Completed | 0 | 0 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Obese (NO): Non obese patients. Patients with a BMI < 29.9 scheduled for clinically indicated laparoscopic abdominal surgery.
- Super-morbidly Obese (SMO): Patients with a BMI > 50.0 scheduled for clinically indicated laparoscopic abdominal surgery.
- Total: Total of all reporting groups
Arm/Group | Non-Obese (NO) | Morbidly Obese (MO) | Super-morbidly Obese (SMO) | Total
Number analyzed (Participants) | 10 | 10 | 30 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Between 18 and 65 years | 10 (0) | 10 (0) | 30 (0) | 50 (0)
  >=65 years | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 16 | 26
  Male | 5 | 5 | 14 | 24

OUTCOME MEASURES:

1. Primary Outcome: Size of Adipocytes
Description: The mean diameters of omental adipocytes were measured
Time Frame: 4 years
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Non-Obese (NO) | Morbidly Obese (MO) | Super-morbidly Obese (SMO)
Number analyzed (Participants) | 10 | 10 | 30
µm | 73.4 (16.1) | 99.0 (24.0) | 103.0 (14.2)

2. Primary Outcome: Maximum Reaction Velocity (Vmax) for Facilitated LCFA Uptake
Description: The Vmax for facilitated Long Chain Fatty Acids (LCFA) uptake by omental adipocytes was measured.
Time Frame: 4 years
Measure: Mean (Standard Deviation); unit: pmol/sec
Arm/Group | Non-Obese (NO) | Morbidly Obese (MO) | Super-morbidly Obese (SMO)
Number analyzed (Participants) | 10 | 10 | 30
pmol/sec | 8.3 (1.8) | 20.9 (4.1) | 68.7 (9.45)

3. Secondary Outcome: Maximum Reaction Velocity (Vmax) for Fatty Acid Uptake Relative to Adipocyte Cell Surface Area
Description: Fatty acid uptake was expressed relative to adipocyte cell surface area [Vmax'(pmol/sec/µm^2) = Vmax/(cell surface area) X 10^8].
Time Frame: 4 years
Measure: Mean (Standard Deviation); unit: pmol/sec/μm^2
Arm/Group | Non-Obese (NO) | Morbidly Obese (MO) | Super-morbidly Obese (SMO)
Number analyzed (Participants) | 10 | 10 | 30
pmol/sec/μm^2 | 0.88 (0.39) | 1.24 (0.36) | 3.21 (1.89)

ADVERSE EVENTS:
Arm/Group | Non-Obese (NO) | Morbidly Obese (MO) | Super-morbidly Obese (SMO)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No